CLINICAL TRIAL: NCT02827968
Title: A Phase I, Open Label, Dose Escalation Study of The Safety and Pharmacokinetics of Anti-PD-L1 Monoclonal Antibody KN035 Administered in Subcutaneous Injection as A Single Agent to Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: Phase 1 Study of Anti-PD-L1 Monoclonal Antibody KN035 to Treat Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 3D Medicines (Sichuan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: 3D Medicines (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN035-US-001
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-03

CONDITIONS: Solid Tumors
Keywords: PDL-1
MeSH Terms: interventions — envafolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KN035 (Experimental): Cohorts of 3-6 subjects will be enrolled sequentially at escalating doses of 1, 2.5, 5 and 10 mg/kg weekly.
  Interventions: Drug: KN035

INTERVENTIONS:
Drug: KN035 — KN035 is a monoclonal antibody drug which is formulated for subcutaneous injection in a single-use vial (brown neutral borosilicate) containing a total of 300 mg antibody in 1.5 ml of solution.

SUMMARY:
This is an open label, dose escalation study to evaluate the safety and tolerability of KN035 in advanced and metastatic solid tumor.

DETAILED DESCRIPTION:
The dose escalation will follow the traditional 3+3 design. Cohorts of 3-6 subjects will be enrolled sequentially at escalating doses of 1, 2.5, 5 and 10 mg/kg weekly. Dosing schedule for cohorts 2 and above may change after interim PK analysis after Cohort 1 Cycle 1 to bi-weekly or other regimen based on elimination profile of KN035 to avoid excessive drug accumulation. Dose escalation will continue until identification of MTD, up to a maximum dose of 10 mg/kg. MTD is defined as the highest dose studied at which no more than 1 of 6 subjects has experienced a dose-limiting toxicity (DLT) in Cycle 1.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histological or cytological diagnosis of any type of carcinoma, progressive metastatic disease, or progressive locally advanced disease not amenable to local therapy. Subjects must have failed established standard medical anti-cancer therapies for a given tumor type or have been intolerant to such therapy, or in the opinion of the Investigator have been considered ineligible for a particular form of standard therapy on medical grounds.
* Subject is male or female and ≥ 18 years of age on day of signing informed consent.
* Subject must have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Subject must have adequate hematologic and organ function. Note: If subject is receiving anticoagulants, then value must be within therapeutic range for the condition the subject is being treated for.
* Subject has voluntarily agreed to participate by giving written informed consent. If subject has agreed to a newly obtained biopsy of tumor (that can be biopsied based on Investigator's assessment). Tissue obtained for the biopsy must not be previously irradiated. No systemic antineoplastic therapy may be received by the subject between the time of the biopsy and the first administration of KN035.
* Female subject of childbearing potential has a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the subject to be eligible.
* Female subjects enrolled in the study, who are not free from menses for > 2 years, post hysterectomy/oophorectomy, or surgically sterilized, must be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy or to abstain from heterosexual activity throughout the study, starting with Visit 1 through 120 days after the last dose of study therapy. Approved contraceptive methods include for example; intra uterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, or female condom with spermicide. Spermicides alone are not an acceptable method of contraception.

Male subjects must agree to use an adequate method of contraception starting with the first dose of study drug through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Subject who not recovered from the effects of any prior chemotherapy, radioactive, or biological cancer therapy prior to the first dose of study therapy (for prior cancer therapy drugs, a washout of 5 half-lives is required), or who has not recovered to CTCAE Grade 1 or better from the adverse events due to cancer therapeutics administered more than 4 weeks earlier. Subject who has had erlotinib, gefitinib, afatinib, or crizotinib within 1 week prior to the first dose of study therapy, or who has not recovered to CTCAE Grade 1 or better from the adverse events due to any of these drugs administered more than 1 week earlier.
* Subject is expected to require any other form of antineoplastic therapy while on study (including maintenance therapy with another agent for NSCLC).
* Subject had prior treatment targeting PD-L1 axis or CTLA 4. Subjects with prior treatment targeting PD-1 are allowed to enroll if the subject has a washout time of at least 4 weeks. Examples of such agents include (but are not limited to): BMS-936559 (MDX 1105); MPDL3280A (RG7446); and MEDI4736.
* Subject has a medical condition that requires chronic systemic steroid therapy or requires any other form of immunosuppressive medication. However, subjects using physiologic replacement doses of hydrocortisone, or its equivalent, will be considered eligible for this study: up to 20 mg hydrocortisone (or 5 mg of prednisone) in the morning and 10 mg hydrocortisone (or 2.5 mg of prednisone) in the evening.
* Subject has risk factors for bowel obstruction or bowel perforation (examples include but not limited to a history of acute diverticulitis, intra-abdominal abscess, or abdominal carcinomatosis).
* Subject has a known history of a hematologic malignancy, malignant primary brain tumor or malignant sarcoma, or of another malignant primary solid tumor, unless the subject has undergone potentially curative therapy with no evidence of that disease for 5 years.

Note: The time requirement does not apply to subjects who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.

* Subject has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks prior to study entry, have no evidence of new or enlarging brain metastases and are off steroids for at least 7 days from first dose of KN035.
* Subject previously had a severe hypersensitivity reaction to treatment with another mAb.
* Subject has a history of pneumonitis or interstitial lung disease.
* Subject has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism that is stable on hormone replacement will not be excluded from the study.
* Subject has an active infection requiring therapy.
* Subject is positive for Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), active hepatitis B (HBsAg reactive) or hepatitis C (HCV RNA (qualitative) is detected); subjects with negative hepatitis C antibody testing may not need RNA testing.
* Subject has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
* Subject has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Subject has a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds (ms)), or a history of additional risk factors for torsade de pointes (TdP, e.g., heart failure, hypokalemia, family history of Long QT Syndrome), or is using concomitant medications that prolong the QT/QTc interval.
* Subject is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
* Subjects with symptomatic ascites or pleural effusion. A subject who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible.
* Subject is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | From screening to up to cycle 1 (28 days)
Percentage of participants with adverse events (AEs), serious adverse events and AEs of special interest | From screening to up to 3 months after the last dose of study drug (up to approximately 2 years)

SECONDARY OUTCOMES:
Serum Concentrations of KN035 | From Pre-dose of the first dose to up to 3 months after the last dose of study drug (up to approximately 2 years)
  Blood samples will be collected at Pre-dose, 6hrs,24 hrs,48hrs,96hrs after the end of the first injection of KN035, after injection of KN035 at Day 8, 15, 22 in first cycle and pre-dose and within 24hrs of following cycles(Cycle length = 28 days), and at the mandatory Safety Follow-up visits
Percentage of Participants with Best Overall Response as determined by Response Evaluation Criteria in Solid Tumours (RECIST) Version (v) 1.1 | Baseline until disease progression, death, loss to follow-up, initiation of another anti-cancer treatment, withdrawal of consent, or study termination by the Sponsor, whichever occurs first (up to approximately 2 years)
Percentage of Participants with Objective Response as determined by RECIST v1.1 | Baseline until disease progression, death, loss to follow-up, initiation of another anti-cancer treatment, withdrawal of consent, or study termination by the Sponsor, whichever occurs first (up to approximately 2 years)
Duration of Objective Response as determined by RECIST v1.1 | Baseline until disease progression, death, loss to follow-up, initiation of another anti-cancer treatment, withdrawal of consent, or study termination by the Sponsor, whichever occurs first (up to approximately 2 years)
Progression Free Survival Duration as determined by RECIST v1.1 | Baseline until disease progression, death, loss to follow-up, initiation of another anti-cancer treatment, withdrawal of consent, or study termination by the Sponsor, whichever occurs first (up to approximately 2 years)
Overall Survival Duration | Baseline until disease progression, death, loss to follow-up, initiation of another anti-cancer treatment, withdrawal of consent, or study termination by the Sponsor, whichever occurs first (up to approximately 2 years)
Percentage of participants with anti-therapeutic antibody (ATA) | From screening to up to 3 months after the last dose of study drug (up to approximately 2 years)
  Blood samples will be collected at Pre-dose of Cycle 1 and D1,8 of the following cycles.

CONTACTS AND LOCATIONS:
Overall Officials: David Liu, M.D., Study Chair — 3D Medicines
Locations (2):
- United States (2):
  - Horizon Oncology Research, INC, Lafayette, Indiana
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Papadopoulos KP, Harb W, Peer CJ, Hua Q, Xu S, Lu H, Lu N, He Y, Xu T, Dong R, Gong J, Liu D. First-in-Human Phase I Study of Envafolimab, a Novel Subcutaneous Single-Domain Anti-PD-L1 Antibody, in Patients with Advanced Solid Tumors. Oncologist. 2021 Sep;26(9):e1514-e1525. doi: 10.1002/onco.13817. Epub 2021 May 27. PMID 33973293